CLINICAL TRIAL: NCT05587673
Title: A Pilot Study Investigating the Feasibility and Efficacy of Locoregional Intra-arterial Administration of Methylprednisolone as a Bridge Therapy to Treat Symptomatic Flares in Inflammatory Bowel Disease
Brief Title: High Dose Steroid Therapy to Treat Flares in Patients With Inflammatory Bowel Disease (IBD)
Acronym: IBDIR
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Avnesh Thakor, Associate Professor of Radiology, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 64154
Record Dates: First submitted 2022-10-14; First posted 2022-10-20 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Inflammatory Bowel Diseases; Crohn Disease; Ulcerative Colitis; Indeterminate Colitis
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative | interventions — Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Methylprednisolone (Experimental): Participants who have failed first line therapy and are still experiencing flare symptoms.
  Interventions: Drug: Methylprednisolone

INTERVENTIONS:
Drug: Methylprednisolone — High dose steroid injected directly into the inflamed bowel segment(s) via its arterial blood supply.

SUMMARY:
This study will examine whether delivery of high dose steroids, directly into the inflamed bowel via its arterial blood supply, will be better for treating uncontrolled flares of inflammatory bowel disease in patients compared to conventional intra-venous or oral administration of this drug. Patients aged 4-25 years of age will be recruited.

In this study, the Investigator hopes to also learn how this directed steroid delivery during an active flare will improve patient symptoms as well as the appearance of inflamed segments of bowel determined by imaging or biopsy (i.e. at the time of endoscopy). Additional data will determine how the blood vessels in the bowel affect, and potentially even drive the mechanisms, of inflammatory bowel disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosis of inflammatory bowel disease (IBD) or patients who have an established diagnosis of IBD and are experiencing an acute flare which is not being controlled with first line therapy
* Patients present with typical IBD symptoms which will include, but are not limited to, abdominal pain, loss of appetite, rectal bleeding, diarrhea, obstruction, or passage of mucus.
* Patients referred by the GI team.
* Patients (or guardians/parents) must be able and willing to give consent (or assent where applicable) and be able to attend all study visits.

Exclusion Criteria:

* Patients with MR unsafe metallic implants that will not be able to undergo the MRI portion of the study.
* Patients with renal function impairment (GFR < 45 mL/min) preventing contrast administration.
* Patients with contrast allergy.

Ages: 4 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2022-10-06 (Actual); Primary Completion 2023-10-11 (Actual); Study Completion 2024-10-11 (Actual)

PRIMARY OUTCOMES:
Number of patients with symptomatic, imaging or biopsy related improvement in their IBD symptoms | Baseline through week 6
  Number of patients who have symptomatic, imaging or biopsy related improvement in their IBD symptoms following locoregional intraarterial methylprednisolone administration into the affected segment of bowel.

SECONDARY OUTCOMES:
Number of patients in which pre-procedural and procedural imaging can be correlated with clinical outcomes following therapy | Month 6
  Patients will have their pre-procedural and procedural imaging correlated with clinical outcomes following therapy.
Number of patients who have molecular changes correlated with improvement in symptoms following intraarterial steroid therapy. | Month 6
  Number of patients who have molecular changes on their pre and post therapy biopsy which can be correlated with improvement in symptoms or imaging data from a patient.

CONTACTS AND LOCATIONS:
Overall Officials: Avnesh Thakor, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No